CLINICAL TRIAL: NCT02314793
Title: A Phase 1 Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP2205 in Healthy Young Males and Females and Elderly Females and to Evaluate the Effect of Food on the Pharmacokinetics of a Single Dose of ASP2205
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of ASP2205 in Healthy Young Males and Females and Elderly Females and to Evaluate the Effect of Food on the Pharmacokinetics of a Single Dose of of ASP2205
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been terminated because of operational reasons.
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2205-CL-0001; 2014-003059-71 (EudraCT Number)
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP2205
Keywords: Pharmacokinetics; ASP2205
MeSH Terms: interventions — ASP2205

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1: Single Ascending Dose ASP2205 (Fasting) (Experimental): Young male and female subjects will receive single doses of ASP2205 in a dose escalation format.
  Interventions: Drug: ASP2205
- Part 1: Single Ascending Dose Placebo (Fasting) (Placebo Comparator): Young male and female subjects will receive single doses of matching placebo in a dose escalation format.
  Interventions: Drug: Placebo
- Part 1: Single Ascending Dose ASP2205 (Fed) (Experimental): Young male and female subjects will receive a single dose of ASP2205
  Interventions: Drug: ASP2205
- Part 2: Multiple Ascending Dose ASP2205, Young females (Experimental): Young female subjects will receive multiple dosing of ASP2205 for 14 days: single doses on days 1 and 14 and depending on the dosing regimen (based on emerging data from Part 1) either once or twice daily dosing from days 2 to 13.
  Interventions: Drug: ASP2205
- Part 2: Multiple Ascending Dose Placebo, Young females (Placebo Comparator): Young female subjects will receive matching placebo for 14 days: single doses on days 1 and 14 and depending on the dosing regimen (based on emerging data from Part 1) either once or twice daily dosing from days 2 to 13.
  Interventions: Drug: Placebo
- Part 2: Multiple Ascending Dose ASP2205, Elderly females (Experimental): Elderly female subjects will receive multiple dosing of ASP2205 for 14 days: single doses on days 1 and 14 and depending on the dosing regimen (based on emerging data from Part 1) either once or twice daily dosing from days 2 to 13.
  Interventions: Drug: ASP2205
- Part 2: Multiple Ascending Dose Placebo, Elderly females (Placebo Comparator): Elderly female subjects will receive matching placebo for 14 days: single doses on days 1 and 14 and depending on the dosing regimen (based on emerging data from Part 1) either once or twice daily dosing from days 2 to 13.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP2205 — oral
  Arms: Part 1: Single Ascending Dose ASP2205 (Fasting); Part 1: Single Ascending Dose ASP2205 (Fed); Part 2: Multiple Ascending Dose ASP2205, Elderly females; Part 2: Multiple Ascending Dose ASP2205, Young females
Drug: Placebo — oral
  Arms: Part 1: Single Ascending Dose Placebo (Fasting); Part 2: Multiple Ascending Dose Placebo, Elderly females; Part 2: Multiple Ascending Dose Placebo, Young females

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending oral doses of ASP2205 in healthy young male and female subjects. This study will also evaluate the safety and tolerability of multiple ascending oral doses of ASP2205 in healthy young and elderly female subjects.

DETAILED DESCRIPTION:
Part 1 is a single ascending dose investigator-blinded study in healthy young male and female subjects. Six doses of ASP2205 or matching placebo will be given to separate cohorts consisting of 8 subjects each, with 6 subjects receiving ASP2205 and 2 subjects receiving matching placebo. ASP2205 or matching placebo will be given as a single oral dose under fasted conditions.

The effect of a high-calorie high-fat meal (breakfast) on the safety, tolerability and pharmacokinetics of a single oral dose of ASP2205 will be evaluated in a separate cohort of 8 subjects in an open-label manner.

Part 2 is a multiple ascending dose subject- and investigator-blinded study comprising 3 cohorts with each 12 healthy young (aged 25 to 55 years) female subjects and 1 cohort with 12 healthy elderly (aged 65 years or older) female subjects who will receive ASP2205 or matching placebo. Nine subjects in each cohort will be treated with ASP2205 and 3 subjects will be treated with matching placebo (ratio 3:1).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy young male or female subject aged 25 to 55 years, inclusive, at screening (part 1 and 2) or healthy elderly female subject aged ≥ 65 years, inclusive, at screening (part 2 only).
* Subject has a body mass index (BMI) range of 18.5 - 30.0 kg/m2, inclusive. The subject weighs at least 50 kg (at screening).
* Subject agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP2205 or any components of the formulations used.
* Subject has any of the liver function tests (LTs; aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase (ALP), gamma glutamyl transferase, total bilirubin [TBL]) above the upper limit of normal (ULN). In such a case, the assessment may be repeated once (admission to the clinical unit).
* Subject has at screening any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies).
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic (including surgical procedures to treat pelvic trauma), pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to admission to the clinical unit.
* Subject has a relevant history of attempted suicide or suicidal behavior. Any recent suicidal ideation within the last 6 months or who are at significant risk to commit suicide.
* Subject has any clinically significant abnormality.
* Subject has a mean pulse < 40 or > 90 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean DBP > 90 mmHg (elderly subjects: mean SBP > 160 mmHg; mean DBP > 100 mmHg) (vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) prior to the admission to the clinical unit (triplicates taken at screening and on admission to the clinical unit). If the mean blood pressure exceeds the limits above, 1 additional triplicate can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) > 430 ms (for male subjects) and > 450 ms (for female subjects) at admission to the clinical unit. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken.
* Subject uses any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day) and except for use of contraceptives or hormone replacement therapy.
* Subject has a history of smoking within 6 months prior to admission to the clinical unit.
* Subject has a history of drinking > 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) (> 14 units of alcohol for female subjects) within 3 months prior to admission to the clinical unit.
* Subject uses grapefruit juice (more than 3 × 200 mL) or products containing grapefruit and/or Seville oranges (more than 3 times) in the week prior to admission to the clinical unit until ESV, as reported by the subject.
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit.
* Subject regularly uses any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit.
* Subject had significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (immunoglobulin M) (anti-HAV [IgM]), hepatitis C virus antibodies (anti-HCV) or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at screening.
* Subject has been treated with any investigational drugs within 90 days or 5 terminal half-lives, whichever is longer, prior to drug administration.
* Subject is unable to communicate, read and understand English, or has any other condition which makes the subject unsuitable for study participation.
* Subject is an employee of the Astellas Group or Clinical Research Organization involved in the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Part 1 and Part 2: Safety assessed by nature, frequency and severity of adverse events | up to 29 days
Part 1 and Part 2: Safety assessed by vital signs | up to 29 days
  Vital signs include blood pressure, pulse rate, body temperature
Part 1 and Part 2: Safety assessed by orthostatic challenge test | up to 29 days
Part 1 and Part 2: Assessment of clinical laboratory tests | up to 29 days
  Clinical laboratory tests include hematology, biochemistry and urinalysis
Part 1 and Part 2: Safety assessed by routine 12 lead electrocardiogram (ECG) | up to 29 days
Part 1 and Part 2: Safety assessed by continuous cardiac monitoring (Holter ECG) | up to 29 days
Part 1: Safety assessed by real-time cardiac monitoring (ECG telemetry) | up to 16 days

SECONDARY OUTCOMES:
Part 1 and Part 2: Safety laboratory test: prolactin | up to 29 days
Part 1 and Part 2: Safety laboratory test: cortisol | up to 29 days
Part 1 and Part 2: Safety laboratory test: bicarbonate (HCO3) | up to 29 days
Part 1 and Part 2: Safety assessed by chemistry profile | up to 29 days
  Chemistry profile includes total cholesterol, high-density lipoprotein (HDL) / low-density lipoprotein (LDL), triglycerides
Part 1 and Part 2: Safety laboratory test: fasting blood glucose | up to 29 days
Part 1 and Part 2: Safety laboratory test: creatinine urine | up to 29 days
Part 1: Central nervous system (CNS) safety monitoring: Bond & Lader visual analogue scale (VAS) | up to 4 days
Part 1: CNS safety monitoring: Drug effects questionnaire (DEQ) VAS | up to 4 days
  PhenX toolkit version
Part 1: Pharmacokinetics profile of ASP2205 in plasma: AUCinf, AUCinf (% extrapolated), AUClast, AUC24, CL/F, Cmax, terminal elimination rate constant, MRT, tlag, tmax, t1/2, Vz/F | Day 1
  Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf), percentage of AUCinf due to extrapolation from tlast to time infinity (AUCinf %extrapolated), AUC from the time of dosing to the last measurable concentration (AUClast), AUC from the time of dosing to 24 hours (AUC24), apparent total systemic clearance after single or multiple extravascular dosing (CL/F), maximum concentration (Cmax), mean residence time (MRT), time prior to the time corresponding to the first measurable (nonzero) concentration (tlag), time to maximum concentration (tmax), terminal elimination half-life (t1/2), apparent volume of distribution during the terminal elimination phase after single or multiple extravascular dosing (Vz/F)
Part 1: Pharmacokinetics profile of ASP2205 in urine: Aeinf, Aeinf%, Aelast, Aelast%, CLR | Day 1
  Cumulative amount of drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf), percentage of drug dose excreted into urine from time of dosing extrapolated to time infinity (Aeinf%), cumulative amount of drug excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast), percentage of drug dose excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast%), renal clearance (CLR)
Part 2: Safety laboratory test: di-docosahexaenoyl-bis(monoacylglycerol) phosphate (di-22:6-BMP) in serum and urine | up to 29 days
Part 2: CNS safety monitoring: CogState's neurocognition test battery (short version) | up to 14 days
Part 2: CNS safety monitoring: Bond & Lader VAS | up to 17 days
Part 2: CNS safety monitoring: DEQ VAS | Time Frame : up to 13 days
  PhenX toolkit version
Part 2: CNS safety monitoring: Addiction Research Center Inventory (49-item short form) (ARCI-49) | up to 13 days
Part 2: CNS safety monitoring: Physician Withdrawal Checklist | up to 29 days
Part 2: CNS safety monitoring: Columbia - Suicide Severity Rate Scale (C-SSRS) | up to 29 days
Part 2: Appetite visual analogue scale (AVAS) | up to 15 days
Part 2: Nausea VAS | up to 15 days
  From the McGill Nausea questionnaire
Part 2: Body weight | up to 29 days
Part 2: Total daily urine production (24-hour volume) | up to 15 days
Part 2: Total daily urine osmolality (24 hour pooled sample from each void) | up to 15 days
Part 2: Total daily fluid intake | up to 15 days
Part 2: Pharmacokinetic profile of ASP2205 in plasma: AUC24, Cmax, tlag, tmax | Day 1
Part 2: Pharmacokinetic parameter: Ctrough | Day 1 immediately prior to dosing (morning Ctrough and, only in case of twice daily dosing, evening C trough): days 2, 4, 6, 8, 10, 12
Part 2: Pharmacokinetic profile of ASP2205 in plasma: AUCtau, Cmax, tmax | Days 12, 13 (in case of twice daily dosing)
Part 2: Pharmacokinetic profile of ASP2205 in plasma: AUCtau, CL/F, Cmax, terminal elimination rate constant, MRT, peak trough ratio (PTR), accumulation ratio calculated using the area under the concentration -time curve [Rac(AUC)], tmax, t1/2, VzF | Day 14
Part 2: Pharmacokinetic profile of ASP2205 in urine: Aetau, Aetau%, CLR | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Site GB44001, Harrow, United Kingdom